CLINICAL TRIAL: NCT07045779
Title: The OMBIT Study: Oral Myofunctional Pattern in Children With Anterior Open Bite
Brief Title: Oral Myofunctional Pattern in Children With Anterior Open Bite
Acronym: OMBIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2022-0135
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Orofacial Myofunctional Disorders; Anterior Open Bite Malocclusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional OMT (Experimental): Participants who are randomly assigned to this arm, will receive traditional orofacial myofunctional therapy (OMT), consisting of interventions targeting orofacial strength, orofacial differentiation, breathing pattern, orofacial resting postures, and swallowing pattern.
  Interventions: Behavioral: Orofacial myofunctional therapy - traditional
- Reduced OMT (Experimental): Participants who are randomly assigned to this arm, will receive reduced orofacial myofunctional therapy (OMT), consisting of interventions targeting orofacial differentiation, breathing pattern, and orofacial resting postures.
  Interventions: Behavioral: Orofacial myofunctional therapy - reduced
- Sham treatment (Sham Comparator): Participants who are randomly assigned to this arm, will receive a sham treatment. This active control intervention will not include any of the exercises included in the experimental treatment arms. The sham treatment program will include exercises from an evidence-based vocal warm up program, with exclusion of the exercises that include active involvement of the tongue or lips. Furthermore, exercises regarding body posture (no focus on articulators), relaxation and voice onset will be included. This sham treatment program will be provided by the same speech-language pathologist with comparable motivation techniques as those applied in the real OMT programs. Patients and parents will initially not be informed about the actual purpose of this sham treatment. A debriefing will take place after the follow-up phase.
  Interventions: Behavioral: Vocal warm up

INTERVENTIONS:
Behavioral: Orofacial myofunctional therapy - traditional — Behavioral interventions, like orofacial myofunctional therapy (OMT), target brain reorganization and plasticity by establishing new motor patterns or re-establishing old ones. The aim of OMT is to correct pathological function and resting positions based on the equilibrium theory. A service model that is often used in OMT is the model provided by Garliner, which includes a 10 week OMT program with a frequency of one session of 45 minutes per week together with home practice. Treatment sessions will be used to introduce and practice new exercises, to monitor home practice and motivation of the patients. Additionally, the participant will be instructed to perform the same exercises from the treatment session at home daily. This intervention will consist of (1) creating awareness, (2) establishing nasal breathing, (3) labial seal and lip closure exercises, (4) tongue posture exercises, (5) lip and tongue strengthening, (6) practicing a physiological swallowing act.
  Arms: Traditional OMT
Behavioral: Orofacial myofunctional therapy - reduced — Behavioral interventions, like orofacial myofunctional therapy (OMT), target brain reorganization and plasticity by establishing new motor patterns or re-establishing old ones. The aim of OMT is to correct pathological function and resting positions based on the equilibrium theory. A service model that is often used in OMT is the model provided by Garliner, which includes a 10 week OMT program with a frequency of one session of 45 minutes per week together with home practice. Treatment sessions will be used to introduce and practice new exercises, to monitor home practice and motivation of the patients. Additionally, the participant will be instructed to perform the same exercises from the treatment session at home daily. This intervention will consist of (1) creating awareness, (2) establishing nasal breathing, (3) labial seal and lip closure exercises, (4) tongue posture exercises.
  Arms: Reduced OMT
Behavioral: Vocal warm up — The sham treatment program will include exercises from an evidence-based vocal warm up program, with exclusion of the exercises that include active involvement of the tongue or lips. Exercises that will be included are: open mouth approach, glottal fry, producing ascending and descending tones and the hand-over-mouth technique. These exercises aim to improve the dynamics of the extrinsic and intrinsic laryngeal muscles and therefore are expected not to interfere with the content of the OMT program. Furthermore, exercises regarding body posture (no focus on articulators), relaxation and voice onset will be included. This sham treatment program will be provided by the same speech-language pathologist with comparable motivation techniques as those applied in the real OMT programs.
  Arms: Sham treatment

SUMMARY:
Oral myofunctional disorders (OMD) are a key, internationally acknowledged environmental factor causing dental and skeletal malocclusion. For the past 15 years, research regarding the efficacy of orofacial myofunctional therapy (OMT) to reduce OMD and to contribute to the treatment of malocclusions has been significantly increased. Despite the growing interest, high-quality evidence is still lacking because studies show a lack of standardized assessment techniques, outcome measures, and inclusion criteria, important methodological limitations such as small sample sizes, a variety of content and service delivery models and a lack of long-term follow-up.

The goal of this clinical trial is to evaluate the effects of structured OMT on anterior open bite (AOB) in children in early or intermediate mixed dentition. The main questions it aims to answer are:

* Does a structured OMT program affect orofacial myofunctional patterns, dental occlusion, and oral health-related quality of life (OHRQoL) in children with AOB?
* Are there differences in treatment outcomes between children receiving a traditional OMT program, a reduced OMT program, and a sham treatment?

Participants will undergo baseline and follow-up assessments of dental occlusion, orofacial myofunctional patterns, and OHRQoL. They will follow a structured OMT protocol tailored to their assigned group and participate in weekly therapy sessions over a defined intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anterior open bite (AOB)
* Early or intermediate mixed dentition phase

Exclusion Criteria:

* History of or active engagement in orofacial myofunctional therapy (OMT)
* History of or active engagement in orthodontic therapy
* Congenital abnormalities, syndromes, or surgical needs affecting the oral and maxillofacial region
* Disorders affecting motor or cognitive development
* Current or recent (< 3 months) non-nutritive sucking habits

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dental occlusion characteristics | From enrollment until 12 months after conclusion of treatment
  Measurement of dental occlusion characteristics (overbite, overjet, palatal surface area, palatal volume) will be based on 3D digital intraoral scans. The chief among which, anterior open bite, will be measured by vertical gap measurement (mm), i.e. the vertical distance between the incisal edge of the maxillary and mandibular central incisors when in occlusion.
Orofacial myofunctional status | From enrollment until 12 months after conclusion of treatment
  Orofacial myofunctional status will be evaluated using the Orofacial Myofunctional Evaluation with Scores (OMES) protocol, a validated measure quantifying orofacial myofunctional behavior (with a lower score indicative of a more impaired orofacial function). Additionally, submandibular ultrasonography will be used to verify tongue posture at rest and swallowing pattern.

SECONDARY OUTCOMES:
Oral health-related quality of life | From enrollment until 12 months after conclusion of treatment
  OHRQoL will be assessed using the Childrens Oral Health Impact Profile (COHIP) (a higher score is indicative of a better OHRQoL).
Orofacial strength | From enrollment until 12 months after conclusion of treatment
  Maximal strength and endurance of tongue and lips will be assessed using the Iowa Oral Performance Instrument (IOPI).

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Ghent; Kim Bettens, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No